CLINICAL TRIAL: NCT04428424
Title: The Impact of RF, and Anti-CCP on RA Patients in Response to Etanercept
Brief Title: Study To Evaluate The Response To Enbrel And The Impact Of Rheumatoid Factor(RF) And Anti-Cyclic Citrullinated Peptide(Anti-CCP) In Rheumatoid Arthritis(RA) Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801417
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with rheumatoid arthritis: Iraqi patients with rheumatoid arthritis that received Enbrel as treatment for disease
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Enbrel — As provided in real world practice

SUMMARY:
This study is to evaluate available local data in Iraqi patients with rheumatoid arthritis on Enbrel treatment with regards to the impact of Rheumatoid factor and Anti-cyclic citrullinated peptide using data from the Baghdad Teaching Hospital registry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed RA patients.

  -≥18 years of age
* Did not receive previous another biological treatment

Exclusion Criteria:

* Had previous biological treatment
* Use of etanercept for less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients data from the local registry at the Baghdad Teaching Hospital registry.
Sampling Method: Non-Probability Sample
Enrollment: 1493 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1801417

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants with rheumatoid arthritis (RA) and who received etanercept from Baghdad Teaching Hospital (Rheumatology center) from May 2012 until August 2019 were included in this study. Their data was collected from the Baghdad Teaching Hospital registry and retrospectively assessed for 1 month.
Period: Overall Study
Arm/Group | Etanercept
Started | 1493
Completed | 1246
Not Completed | 247
Not completed — Does not meet entrance criteria | 132
Not completed — Lost to Follow-up | 115

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants who were included in this study.
Groups:
- Etanercept: Participants with RA and who received etanercept from Baghdad Teaching Hospital (Rheumatology center) from May 2012 until August 2019 were included in this study. Their data was collected from the Baghdad Teaching Hospital registry and retrospectively assessed for 1 month.
Arm/Group | Etanercept
Number analyzed (Participants) | 1493
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1234
  Male | 259
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score 28 (DAS28) in Participants With Positive Rheumatoid Factor (RF) and Anti-Cyclic Citrullinated Peptide (ACCP) at Last Follow-up Visit (Month 12)
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (in millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated high disease activity). DAS28 less than equal to (<=) 3.2 = low disease activity, DAS28 greater than (>) 3.2 to 5.1 = moderate to high disease activity. DAS28 score in participants with positive RF and ACCP were reported in this outcome measure.
Time Frame: Month 12 visit during retrospective data collection period of approximately 7 years
Population: Analysis was performed on all participants who were included in this study. Here "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for this outcome measure for specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1122
units on a scale
  Positive RF | 3.13 (1.6)
  Positive ACCP: number analyzed (Participants) | 1054
  Positive ACCP | 3.1 (1.58)

2. Primary Outcome: Clinical Disease Activity Index (CDAI) Score in Participants With Positive Rheumatoid Factor (RF) and Anti-Cyclic Citrullinated Peptide (ACCP) at Last Follow-up Visit (Month 12)
Description: The CDAI is the numerical sum of 4 outcome parameters: tender joint count (TJC) and SJC based on a 28-joint assessment, PGA and physician global assessment (PhGA) assessed on 0 to 10 centimeter (cm) visual analog scale (VAS); higher scores = high disease activity. CDAI total score = 0 to 76. CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, > 10 to 22 = moderate disease activity and > 22 = high disease activity. CDAI score in participants with positive RF and ACCP were reported in this outcome measure.
Time Frame: Month 12 visit during retrospective data collection period of approximately 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 1122
units on a scale
  Positive RF | 8.0 (10.4)
  Positive ACCP: number analyzed (Participants) | 1054
  Positive ACCP | 8.2 (10.9)

3. Primary Outcome: Disease Activity Score 28 (DAS28) in Participants With Negative Rheumatoid Factor (RF) and Anti-Cyclic Citrullinated Peptide (ACCP) at Last Follow-up Visit (Month 12)
Description: DAS28 calculated from the SJC and PJC using the 28 joints count, the ESR (in mm/hour) and PGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated high disease activity). DAS28 <= 3.2 = low disease activity, DAS28 > 3.2 to 5.1 = moderate to high disease activity. DAS28 score in participants with negative RF and ACCP were reported in this outcome measure.
Time Frame: Month 12 visit during retrospective data collection period of approximately 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 439
units on a scale
  Negative RF: number analyzed (Participants) | 371
  Negative RF | 3.10 (1.59)
  Negative ACCP | 3.16 (1.6)

4. Primary Outcome: Clinical Disease Activity Index (CDAI) Score in Participants With Negative Rheumatoid Factor (RF) and Anti-Cyclic Citrullinated Peptide (ACCP) at Last Follow-up Visit (Month 12)
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA and PhGA assessed on 0 to 10 cm VAS; higher scores = high disease activity. CDAI total score = 0 to 76. CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, > 10 to 22 = moderate disease activity and > 22 = high disease activity. CDAI score in participants with negative RF and ACCP were reported in this outcome measure.
Time Frame: Month 12 visit during retrospective data collection period of approximately 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 439
units on a scale
  Negative RF: number analyzed (Participants) | 371
  Negative RF | 7.3 (9.0)
  Negative ACCP | 6.8 (7.5)

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events not collected during the study
Description: Study involved data that existed as structured data by time of study start. Since, individual participant data were not retrieved or validated, it was not possible to link (i.e. identify a potential association between) a particular product and medical event for any individual. Thus, minimum criteria for reporting an adverse event (i.e. identifiable participant, identifiable reporter, a suspect product, and event) was not met, hence, safety data was not planned to be collected and reported.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT04428424/Prot_SAP_000.pdf